CLINICAL TRIAL: NCT05567393
Title: A Randomized, Double-blind, Placebo-Controlled, Three-part Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-951 in Healthy Subjects
Brief Title: A Study of TAK-951 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-951-1001
Record Dates: First submitted 2021-10-25; First posted 2022-10-05 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part 1 (SRD): Pooled Placebo (Placebo Comparator): TAK-951 placebo-matching, single dose, subcutaneous (SC) injection, on Day 1 in fasted healthy participants in the single-rising dose (SRD) period.
  Interventions: Drug: TAK-951 Placebo
- Part 1 (SRD): Cohort 2: TAK-951 Dose 1 (Experimental): TAK-951 Dose 1, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 1: TAK-951 Dose 2 (Experimental): TAK-951 Dose 2, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 15: TAK-951 Dose 2 (Experimental): TAK-951 Dose 2, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 3: TAK-951 Dose 3 (Experimental): TAK-951 Dose 3, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 4: TAK-951 Dose 4 (Experimental): TAK-951 Dose 4, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 5: TAK-951 Dose 5 (Experimental): TAK-951 Dose 5, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 6: TAK-951 Dose 6 (Experimental): TAK-951 Dose 6, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 13: TAK-951 Dose 7 (Experimental): TAK-951 Dose 7, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 14: TAK-951 Dose 8 (Experimental): TAK-951 Dose 8, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 16: TAK-951 Dose 9 (Experimental): TAK-951 Dose 9, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 17: TAK-951 Dose 10 (Experimental): TAK-951 Dose 10, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 1 (SRD): Cohort 18: TAK-951 Dose 11 (Experimental): TAK-951 Dose 11, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-951
- Part 3 (MRD): Pooled Placebo (Placebo Comparator): TAK-951 placebo-matching, SC injection, for 5 days from Days 1 to 5 in fasted healthy participants in the multiple-rising dose (MRD) period.
  Interventions: Drug: TAK-951 Placebo
- Part 3 (MRD): Cohort 10: TAK-951 Dose 1A (Experimental): TAK-951 Dose 1A, SC injection, for 5 days from Days 1 to 5 in fasted healthy participants in the MRD period.
  Interventions: Drug: TAK-951
- Part 3 (MRD): Cohort 11: TAK-951 Dose 2A (Experimental): TAK-951 Dose 2A, SC injection, for 5 days from Days 1 to 5 in fasted healthy participants in the MRD period.
  Interventions: Drug: TAK-951
- Part 3 (MRD): Cohort 12: TAK-951 Dose 3A (Experimental): TAK-951 Dose 3A, SC injection, for 5 days from Days 1 to 5 in fasted healthy participants in the MRD period.
  Interventions: Drug: TAK-951
- Part 3 (MRD): Cohort 20: TAK-951 Dose 4A (Experimental): TAK-951 Dose 4A, SC injection, for 5 days from Days 1 to 5 in fasted healthy participants in the MRD period.
  Interventions: Drug: TAK-951

INTERVENTIONS:
Drug: TAK-951 Placebo — TAK-951 placebo-matching SC injection
  Arms: Part 1 (SRD): Pooled Placebo; Part 3 (MRD): Pooled Placebo
Drug: TAK-951 — TAK-951 SC injection
  Arms: Part 1 (SRD): Cohort 13: TAK-951 Dose 7; Part 1 (SRD): Cohort 14: TAK-951 Dose 8; Part 1 (SRD): Cohort 15: TAK-951 Dose 2; Part 1 (SRD): Cohort 16: TAK-951 Dose 9; Part 1 (SRD): Cohort 17: TAK-951 Dose 10; Part 1 (SRD): Cohort 18: TAK-951 Dose 11; Part 1 (SRD): Cohort 1: TAK-951 Dose 2; Part 1 (SRD): Cohort 2: TAK-951 Dose 1; Part 1 (SRD): Cohort 3: TAK-951 Dose 3; Part 1 (SRD): Cohort 4: TAK-951 Dose 4; Part 1 (SRD): Cohort 5: TAK-951 Dose 5; Part 1 (SRD): Cohort 6: TAK-951 Dose 6; Part 3 (MRD): Cohort 10: TAK-951 Dose 1A; Part 3 (MRD): Cohort 11: TAK-951 Dose 2A; Part 3 (MRD): Cohort 12: TAK-951 Dose 3A; Part 3 (MRD): Cohort 20: TAK-951 Dose 4A

SUMMARY:
This is a study of TAK-951 for people with symptoms of nausea and vomiting. The main aims of this study in healthy adults are as follows:

* To check for side effects from TAK-951 when given at a slow and fast infusion rate.
* To learn how much TAK-951 participants can receive without getting side effects from it.
* To check how much TAK-951 stays in the blood over time to work out the best dose.

Participants will receive a single infusion of either TAK-951 or placebo. In this study, a placebo looks like TAK-951 but does not have any medicine in it. Participants will receive either a low dose or high dose of TAK-951. The infusion will take from 1-3 hours.

Participants will stay in the study clinic for about 4 days to receive the study medicine (TAK-951 or placebo) and check for side effects. They will have follow-up visits at the clinic about 2 weeks and 4 weeks after treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-951. The study evaluated the safety, tolerability and pharmacokinetics (PK) of TAK-951 in healthy participants.

The study enrolled 128 healthy participants and consisted of 2 parts: Single-rising Dose (SRD) part (13 cohorts) of sequential panel design, and Multiple-rising Dose (MRD) part (5 cohorts) of sequential panel design. Participants in each cohort were randomized to receive treatment with TAK-951 or matching placebo using SC injection, once daily on Day 1 (for SRD part) and twice daily (BID) on Days 1 through 5 (for MRD part) following a minimum fast of 8 hours.

This single center trial was conducted in the United States. The overall time to participate in this study was approximately 155 days.

ELIGIBILITY:
Inclusion Criteria:

1. Have a body mass index (BMI) ≥18 and ≤30.0 (kg/m^2) at the Screening Visit.

Exclusion Criteria:

1. The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency antibody/antigen, at the Screening Visit. Note: Participants with positive hepatitis B virus or hepatitis C virus serology may be enrolled if quantitative polymerase chain reaction for hepatitis B virus or hepatitis C virus ribonucleic acid is negative.
2. The participant had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks before the Screening Visit.
3. Heavy consumption of alcohol within 3 months before screening (>7 drinks/week for women, >14 drinks/week for men, where 1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) or use of soft drugs (such as marijuana) within 3 months before screening, or hard drugs (such as cocaine and phencyclidine) within 1 year before Screening.
4. The participant has used nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 28 days before check-in (Day -1) or cotinine test is positive at Screening or Day -1.
5. The participant has had 3 incidences of vasovagal syncope within the last 5 years.
6. The participant has Brugada syndrome (right bundle branch block [RBBB] pattern with ST-elevation in leads V1-V3).
7. The participant has an average semirecumbent systolic blood pressure <90 millimeters of mercury (mm Hg) or diastolic blood pressure <60 mm Hg at Screening or admission.
8. The participant has an average heart rate (HR) <60 or >100 beats per minute (bpm) [at Screening, at Day -1, or at predose]; athletic participants with an average HR <60 bpm can be enrolled only with medical monitor approval.
9. The participant has orthostatic hypotension defined as a decrease in systolic blood pressure ≥20 mm Hg or a decrease in diastolic blood pressure ≥10 mm Hg after 2 minutes of standing when compared with blood pressure from the sitting position at Screening, and at Day -1. Participants with postural orthostatic tachycardia, defined as HR >120 bpm standing, will also be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment? commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/70abfd11a4c846d2?idFilter=%5B%22TAK-951-1001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 07 March 2019 to 02 November 2020.
Pre-assignment Details: Healthy participants were enrolled into Part 1 and Part 3 of this study. Participants were randomized into 12 cohorts in Part 1 to receive single-rising dose (SRD) and into 4 cohorts in Part 3 to receive multiple-rising doses (MRD) of TAK-951 or matching placebo in a 3:1 ratio. The randomization in Part 3 was based on the safe and tolerable doses determined in Part 1. As pre-specified in the protocol, Part 2 of the study was not conducted.
Groups:
- Part 3 (MRD): Pooled Placebo: TAK-951 placebo-matching, SC injection, for 5 days from Days 1 to 5 in fasted healthy participants in the MRD period.
Period: Overall Study
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Started | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Completed | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all randomized participants who received at least 1 dose of investigational products in each part of the study.
Groups:
- Part 1 (SRD): Pooled Placebo: TAK-951 placebo-matching, single dose, SC injection, on Day 1 in fasted healthy participants in the SRD period.
- Total: Total of all reporting groups
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A | Total
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 128
Age, Continuous [Mean (Full Range); unit: years] | 39.4 [21 to 53] | 35.2 [24 to 42] | 40.0 [28 to 48] | 35.5 [26 to 41] | 41.8 [21 to 52] | 35.2 [23 to 53] | 34.8 [24 to 48] | 32.0 [24 to 43] | 38.7 [28 to 50] | 42.2 [27 to 52] | 34.5 [26 to 49] | 27.8 [20 to 37] | 43.0 [30 to 53] | 37.3 [27 to 48] | 35.2 [27 to 44] | 33.2 [23 to 39] | 41.3 [36 to 48] | 40.3 [31 to 52] | 37.4 [20 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 11
  Male | 21 | 5 | 6 | 5 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 7 | 5 | 5 | 6 | 6 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 0 | 4 | 2 | 36
  Not Hispanic or Latino | 18 | 6 | 5 | 5 | 5 | 4 | 6 | 5 | 4 | 3 | 3 | 4 | 3 | 4 | 4 | 6 | 2 | 4 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 2 | 2 | 2 | 2 | 0 | 2 | 2 | 2 | 0 | 1 | 2 | 1 | 4 | 2 | 1 | 0 | 3 | 41
  White | 9 | 2 | 3 | 4 | 3 | 4 | 3 | 3 | 3 | 5 | 3 | 3 | 5 | 4 | 3 | 4 | 5 | 3 | 69
  More than one race | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 128
Weight [Mean (Full Range); unit: kg] | 81.20 [59.8 to 106.7] | 78.88 [68.4 to 87.8] | 81.45 [64.1 to 96.2] | 74.10 [65.4 to 90.8] | 73.27 [55.4 to 88.9] | 76.65 [64.1 to 93.6] | 80.02 [60.9 to 107.1] | 76.27 [60.2 to 86.0] | 81.27 [76.2 to 86.5] | 78.87 [65.0 to 87.6] | 77.88 [66.1 to 87.5] | 75.17 [57.1 to 86.5] | 74.92 [59.8 to 88.1] | 78.64 [61.8 to 95.0] | 77.68 [65.0 to 88.8] | 76.35 [64.9 to 93.0] | 75.73 [61.5 to 93.1] | 83.75 [71.3 to 97.8] | 77.89 [55.4 to 107.1]
Height [Mean (Full Range); unit: cm] | 176.8 [162 to 195] | 174.3 [170 to 183] | 175.7 [170 to 184] | 177.8 [161 to 184] | 174.5 [164 to 194] | 177.2 [170 to 183] | 182.5 [174 to 193] | 173.8 [169 to 185] | 175.5 [173 to 182] | 174.0 [162 to 186] | 174.0 [158 to 179] | 172.5 [167 to 176] | 175.8 [165 to 189] | 175.3 [158 to 194] | 172.0 [162 to 181] | 174.7 [163 to 185] | 169.3 [160 to 179] | 175.0 [166 to 181] | 175.04 [158 to 195]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — BMI=weight (kg) / [height (m)]^2
  kg/m^2 | 25.99 [20.7 to 30.2] | 26.08 [21.2 to 30.4] | 26.32 [22.2 to 29.3] | 23.43 [19.7 to 26.8] | 23.90 [20.3 to 27.0] | 24.42 [21.5 to 29.9] | 23.88 [18.2 to 28.8] | 25.23 [20.8 to 28.7] | 26.43 [23.7 to 28.6] | 26.07 [20.7 to 28.6] | 25.77 [20.9 to 27.6] | 25.20 [18.9 to 28.0] | 24.25 [21.2 to 30.3] | 25.68 [19.9 to 29.8] | 26.17 [24.8 to 28.3] | 25.00 [21.8 to 29.0] | 26.32 [24.0 to 29.1] | 27.27 [24.8 to 30.2] | 25.41 [18.2 to 30.4]

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 3: Percentage of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included the examination of the abdomen; extremities; head, eyes, ears, nose (HEENT); neurological; skin and mucosae; thorax.
Time Frame: From the first dose of study drug up to follow-up or early termination (Up to approximately 32 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Parts 1 and 3: Percentage of Participants With Markedly Abnormal Values of Vital Signs Parameters
Description: The criteria for markedly abnormal values of vital signs' parameters were: Pulse Rate (beats/minute) <50 and >120; Systolic Blood Pressure [millimeters of mercury (mmHg)] <85 and >180; Diastolic Blood Pressure (mmHg) <50 and >110; Temperature [degrees Celsius (C)] <35.6 and >37.7. Only categories with atleast one participant with events are reported.
Time Frame: From the first dose of study drug up to follow-up or early termination (Up to approximately 32 days)
Population: Safety Set included all randomized participants who received at least 1 dose of investigational products in each part of the study. The values are rounded off to the nearest whole number.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants
  Diastolic Blood Pressure (mmHg) <50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 16.7 | 33.3 | 16.7 | 16.7 | 16.7 | 0 | 0 | 16.7 | 0 | 0
  Pulse Rate (beats/minute) <50 | 8.3 | 16.7 | 0 | 16.7 | 16.7 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50.0 | 50.0 | 50.0 | 0 | 33.3
  Pulse Rate (beats/minute) >120 | 0 | 0 | 0 | 0 | 0 | 0 | 33.3 | 0 | 16.7 | 16.7 | 50.0 | 50.0 | 16.7 | 0 | 0 | 50.0 | 16.7 | 16.7
  Systolic Blood Pressure (mmHg) <85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 33.3 | 16.7 | 16.7 | 0 | 12.5 | 0 | 33.3 | 0 | 0
  Temperature (C) <35.6 | 4.2 | 33.3 | 16.7 | 0 | 16.7 | 16.7 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 16.7 | 25.0 | 33.3 | 16.7 | 16.7 | 16.7

3. Primary Outcome: Parts 1 and 3: Percentage of Participants With Markedly Abnormal Values of 12-Lead Electrocardiogram (ECG) Parameters
Description: The criteria for markedly abnormal values of 12-lead ECG parameters were: ECG Mean Heart Rate (beats/min) <50 beats per minute and >120 beats per minute; PR Interval, Aggregate [milliseconds (msec)] <=80 msec and >=200 msec; QRS Duration, Aggregate (msec) <=80 msec and >=120 msec; QT Interval with Fridericia Correction Method (QTcF) Interval, Aggregate (msec) >=500 msec or >=30 msec change from Baseline and >=450 msec. Only categories with atleast one participant with event are reported.
Time Frame: From the first dose of study drug up to follow-up or early termination (Up to approximately 32 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants
  ECG Mean Heart Rate (beats/minute) <50 | 8.3 | 0 | 0 | 16.7 | 16.7 | 33.3 | 0 | 16.7 | 16.7 | 0 | 16.7 | 16.7 | 0 | 37.5 | 0 | 33.3 | 0 | 16.7
  PR Interval, Aggregate (msec) >=200 | 4.2 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0
  QRS Duration, Aggregate (msec) <=80 | 20.8 | 16.7 | 16.7 | 16.7 | 16.7 | 0 | 33.3 | 16.7 | 0 | 16.7 | 16.7 | 16.7 | 16.7 | 0 | 0 | 33.3 | 16.7 | 16.7

4. Primary Outcome: Parts 1 and 3: Percentage of Participants With Markedly Abnormal Values of Laboratory Parameters
Description: The laboratory parameters of chemistry, and hematology were assessed. Clinical laboratory tests included serum chemistry, hematology, and urinalysis. MAV criteria: Alanine aminotransferase(U/L) >3xupper limit of normal(ULN); Albumin<2.5g/dL,<25g/L; Alkaline phosphatase (U/L)>3 x ULN; Aspartate aminotransferase (U/L)>3 x ULN; Bilirubin>1.5mg/dL, >34.2 µmol/L; Calcium<8.0 mg/dL,LLN-<2.0mmol/L, >1.0mmol/L; Carbon dioxide <8.0 (mmol/L); Chloride<75 mmol/L,>126 mmol/L; Creatinine>177µmol/L; Gamma glutamyl transferase (U/L)>2.0 mg/dL, >3.0 x ULN; Glucose<3 mmol/L,>10 mmol/L; Potassium<3.0 mmol/L >5.5 mmol/L; Protein(g/L)<0.8 x LLN >1.2 x ULN; Sodium<130mmol/L >150mmol/L; Urea nitrogen >10.7; Erythrocytes 10^12erythrocytes/L) <0.8 x LLN,>1.2 x ULN; Hematocrit(%) <0.8 x LLN,>1.2xULN; Hemoglobin(g/L)<0.8 x LLN, >1.2 x ULN; Leukocytes(10^9 leukocytes/L)<0.5 x LLN >1.5 x ULN; platelets(10^9 platelets/L)<75->600. Only categories with atleast one participant with event are reported.
Time Frame: From the first dose of study drug up to follow-up or early termination (Up to approximately 32 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants
  Calcium(mmol/L):Corrected Serum Calcium <LLN 8.0mg/dL;<LLN 2.0mmol/L;Ionized calcium<LLN 1.0mmol/L | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0
  Glucose (mmol/L) >10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0
  Urea Nitrogen (mmol/L) >10.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0

5. Primary Outcome: Parts 1 and 3: Percentage of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug.
Time Frame: From the first dose of study drug up to follow-up or early termination (Up to approximately 32 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants | 16.7 | 16.7 | 16.7 | 16.7 | 16.7 | 16.7 | 33.3 | 50.0 | 50.0 | 83.3 | 66.7 | 83.3 | 33.3 | 37.5 | 16.7 | 83.3 | 66.7 | 83.3

6. Primary Outcome: Parts 1 and 3: Percentage of Participants With Positive Immunogenicity (ADA) Status
Time Frame: From the first dose of study drug up to follow-up or early termination (Up to approximately 32 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 24 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0

7. Secondary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for TAK-951
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Part 1
Population: Part 1: Pharmacokinetic (PK) Set included all participants who received TAK-951 and had at least 1 measurable plasma concentration of TAK-951 in Part 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliters (pg/mL)
Arm/Group | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
picograms per milliliters (pg/mL) | 177 (22.3) | 213 (35.4) | 420 (14.4) | 383 (20.0) | 717 (29.0) | 2070 (24.7) | 3010 (38.4) | 4230 (32.4) | 8920 (41.7) | 8540 (23.6) | 27900 (19.3) | 54300 (14.1)

8. Secondary Outcome: Part 1: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-951
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose in Part 1
Population: PK Set (Part 1) included all participants who received TAK-951 and had at least 1 measurable plasma concentration of TAK-951 in Part 1. Two participants were excluded from the overall number analyzed from 'Part 1 (SRD): Cohort 6: TAK-951 Dose 6' arm as their values were derived from poorly estimated elimination phase during the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms*hour per milliliters(pg*hr/mL)
Arm/Group | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11
Number analyzed (Participants) | 6 | 0 | 6 | 0 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 6
picograms*hour per milliliters(pg*hr/mL) | 813 (14.6) |  | 1960 (8.50) |  | 3920 (12.3) | 9230 (25.7) | 15300 (14.0) | 21700 (34.4) | 46700 (23.3) | 50700 (25.7) | 140000 (17.8) | 340000 (20.8)

9. Secondary Outcome: Part 3: Cmax: Maximum Observed Plasma Concentration for TAK-951 on Day 1
Time Frame: Pre-dose and at multiple time points (up to 24 hours) post-dose on Day 1 in Part 3
Population: PK Set (Part 3) included all participants who received TAK-951 and had at least 1 measurable plasma concentration of TAK-951 in Part 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 6 | 6 | 6 | 6
pg/mL | 1260 (27.1) | 6010 (18.2) | 22400 (25.8) | 33700 (24.6)

10. Secondary Outcome: Part 3: AUCτ: Area Under the Plasma Concentration-time Curve During a Dosing Interval Tau (τ), From Time of First Daily Dose to 8 Hours for TAK-951 on Day 1
Time Frame: Pre-dose and at multiple time points (up to 24 hours) post-dose on Day 1 in Part 3
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
Number analyzed (Participants) | 6 | 6 | 6 | 6
pg*hr/mL | 5420 (25.2) | 25000 (15.9) | 98100 (22.8) | 152000 (29.4)

ADVERSE EVENTS:
Time Frame: From first dose of study drug and up to 30 days post last dose (Parts 1 and 3: Up to approximately 32 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 (SRD): Pooled Placebo | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 | Part 3 (MRD): Pooled Placebo | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/24 | 1/6 | 1/6 | 1/6 | 1/6 | 1/6 | 2/6 | 3/6 | 3/6 | 5/6 | 4/6 | 5/6 | 2/6 | 3/8 | 1/6 | 5/6 | 4/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (SRD): Pooled Placebo (N=24) | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 (N=6) | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 (N=6) | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 (N=6) | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 (N=6) | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 (N=6) | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 (N=6) | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 (N=6) | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 (N=6) | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 (N=6) | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 (N=6) | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 (N=6) | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 (N=6) | Part 3 (MRD): Pooled Placebo (N=8) | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A (N=6) | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A (N=6) | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A (N=6) | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A (N=6)
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (SRD): Pooled Placebo (N=24) | Part 1 (SRD): Cohort 2: TAK-951 Dose 1 (N=6) | Part 1 (SRD): Cohort 1: TAK-951 Dose 2 (N=6) | Part 1 (SRD): Cohort 15: TAK-951 Dose 2 (N=6) | Part 1 (SRD): Cohort 3: TAK-951 Dose 3 (N=6) | Part 1 (SRD): Cohort 4: TAK-951 Dose 4 (N=6) | Part 1 (SRD): Cohort 5: TAK-951 Dose 5 (N=6) | Part 1 (SRD): Cohort 6: TAK-951 Dose 6 (N=6) | Part 1 (SRD): Cohort 13: TAK-951 Dose 7 (N=6) | Part 1 (SRD): Cohort 14: TAK-951 Dose 8 (N=6) | Part 1 (SRD): Cohort 16: TAK-951 Dose 9 (N=6) | Part 1 (SRD): Cohort 17: TAK-951 Dose 10 (N=6) | Part 1 (SRD): Cohort 18: TAK-951 Dose 11 (N=6) | Part 3 (MRD): Pooled Placebo (N=8) | Part 3 (MRD): Cohort 10: TAK-951 Dose 1A (N=6) | Part 3 (MRD): Cohort 11: TAK-951 Dose 2A (N=6) | Part 3 (MRD): Cohort 12: TAK-951 Dose 3A (N=6) | Part 3 (MRD): Cohort 20: TAK-951 Dose 4A (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accelerated idioventricular rhythm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 2 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT05567393/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT05567393/SAP_001.pdf